CLINICAL TRIAL: NCT01658904
Title: Phase I / II Study Of Carfilzomib (CFZ) Intensification Early After Autologous Transplantation (AHCT) For Plasma Cell Myeloma
Brief Title: Carfilzomib and Stem Cell Transplant for Plasma Cell Myeloma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: study closed prematurely because investigator left National Institutes of Health
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daniel Fowler, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120179; 12-C-0179
Record Dates: First submitted 2012-08-03; First posted 2012-08-07 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-04

CONDITIONS: Multiple Myeloma; Leukemia, Plasma Cell
Keywords: Autologous Transplant; Proteasome Inhibitor; Melphalan; Filgrastim
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell | interventions — carfilzomib; Melphalan; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort 1- CFZ 20 mg/m^2 (Day 1,2) (Experimental): Phase I/II study on the backbone of high-dose melphalan on day -2 pre-autologous hematopoietic cell transplantation (AHCT)
  •Addition of an increasing number of doses of Carfilzomib (CFZ) in the early post-AHCT period introduced in a step-wise fashion in 3 successive cohorts of 3 to 15 subjects:
  Cohort 1: add CFZ 20 mg/m^2 intravenous (IV) on days +1, +2
  Cohort 2 : add CFZ 20 mg/m^2 IV on days: +1, +2, +8, +9
  Cohort 3: add CFZ 20 mg/m^2 IV on days: +1, +2, +8, +9 and add an early post-AHCT consolidation following engraftment: CFZ 20 mg/m^2 IV given on days 42-43 then CFZ 56 mg/m^2 IV given on days 49-50, 56-57, then on days 70.
  Interventions: Drug: Carfilzomib; Drug: Melphalan; Drug: Filgrastim
- Cohort 2- CFZ 20 mg/m^2 (Day 1,2,8,9) (Experimental): Phase I/II study on the backbone of high-dose melphalan on day -2 pre-autologous hematopoietic cell transplantation (AHCT)
  •Addition of an increasing number of doses of Carfilzomib (CFZ) in the early post-AHCT period introduced in a step-wise fashion in 3 successive cohorts of 3 to 15 subjects:
  Cohort 1: add CFZ 20 mg/m^2 intravenous (IV) on days +1, +2
  Cohort 2 : add CFZ 20 mg/m^2 IV on days: +1, +2, +8, +9
  Cohort 3: add CFZ 20 mg/m^2 IV on days: +1, +2, +8, +9 and add an early post-AHCT consolidation following engraftment: CFZ 20 mg/m^2 IV given on days 42-43 then CFZ 56 mg/m^2 IV given on days 49-50, 56-57, then on days 70.
  Interventions: Drug: Carfilzomib; Drug: Melphalan; Drug: Filgrastim
- Cohort 3-CFZ 20 mg/m^2 (Day1,2,8,9/AHCT) (Experimental): Phase I/II study on the backbone of high-dose melphalan on day -2 pre-autologous hematopoietic cell transplantation (AHCT)
  •Addition of an increasing number of doses of Carfilzomib (CFZ) in the early post-AHCT period introduced in a step-wise fashion in 3 successive cohorts of 3 to 15 subjects:
  Cohort 1: add CFZ 20 mg/m^2 intravenous (IV) on days +1, +2
  Cohort 2 : add CFZ 20 mg/m^2 IV on days: +1, +2, +8, +9
  Cohort 3: add CFZ 20 mg/m^2 IV on days: +1, +2, +8, +9 and add an early post-AHCT consolidation following engraftment: CFZ 20 mg/m^2 IV given on days 42-43 then CFZ 56 mg/m^2 IV given on days 49-50, 56-57, then on days 70.
  Interventions: Drug: Carfilzomib; Drug: Melphalan; Drug: Filgrastim

INTERVENTIONS:
Drug: Carfilzomib
Drug: Melphalan
Drug: Filgrastim

SUMMARY:
Background:

- Plasma cell myeloma is a type of cancer that affects the plasma cells in the bone marrow. It can be difficult to treat with chemotherapy. One possible treatment combines chemotherapy with a stem cell transplant. To make this treatment more effective, researchers want to give another drug along with the transplant. This drug, carfilzomib, is often used to help treat plasma cell myeloma. However, it is not usually given along with the transplant. Researchers want to see if it is safe and effective to combine the stem cell transplant with carfilzomib, and if it improves the results of the transplant.

Objectives:

- To test the safety and effectiveness of carfilzomib given with stem cell transplant for plasma cell myeloma.

Eligibility:

- Individuals between 18 and 75 years of age who are having a stem cell transplant to treat plasma cell myeloma.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. Imaging studies and a bone marrow biopsy will also be performed.
* Participants will have their own stem cells collected for the transplant. The transplant will be performed according to the standard of care.
* All participants will receive carfilzomib on the first 2 days after transplant. The study doctors will determine the number of additional doses that they may have.
* Treatment will be monitored with frequent blood tests and imaging studies.

DETAILED DESCRIPTION:
Background:

* Despite very significant progress in therapy for plasma cell myeloma (PCM) in the last decade, the disease remains mostly incurable.
* High-dose chemotherapy followed by autologous hematopoietic cell transplantation (AHCT) continues to be a critical component of early treatment for PCM, but it is clear that the disease is not eradicated by the present high-dose therapy strategy, while intensifying the preparative regimen has, to this day, resulted in either no improvement in disease control or increased toxicity.
* Carfilzomib (CFZ) is a newer proteasome inhibitor with increased activity and a safer toxicity profile than bortezomib in PCM. The favorable toxicity profile makes it a likely candidate for increasing anti-PCM drug exposure in the early post-AHCT period.

Objectives:

Primary Objectives

-Evaluate feasibility and toxicity of an increasing number of doses of CFZ administered in the early period post-AHCT for PCM

Secondary Objective

* Evaluate the immune reconstitution post-AHCT following CFZ therapy
* Evaluate the effects of the addition of CFZ in the early post-AHCT period on the response rate at day 100 post-AHCT

Eligibility:

* Newly diagnosed subjects with PCM following induction therapy
* Subjects with documentation of persistent/refractory disease who have received no more than 2 salvage regimens following relapse and who have not undergone AHCT
* Adequate organ functions with no major co-morbidity
* Age greater than 18 years and less than or equal to 75 years

Design:

* Phase I/II study on the backbone of high-dose melphalan on day -2 pre-AHCT
* Addition of an increasing number of doses of CFZ in the early post-AHCT period introduced in a step-wise fashion in 3 successive cohorts of 3 to 15 subjects:

Cohort 1: add CFZ 20 mg/m^2 on days +1, +2

Cohort 2 : add CFZ 20 mg/m^2 on days: +1, +2, +8, +9

Cohort 3: add CFZ 20 mg/m^2 on days: +1, +2, +8, +9 and add an early post-AHCT consolidation following

engraftment: CFZ 20 mg/m^2 given on days 42-43 then CFZ 56 mg/m^2 given on days 49-50, 56-57, then on days 70-71, 77-78 and 84-85

-Dose-limiting toxicity, incidence of engraftment failure and treatment-related mortality are the objects of early stopping rules for safety purposes

ELIGIBILITY:
* INCLUSION CRITERIA:

Multiple myeloma criteria for newly or recently diagnosed subjects

* Presence of clonal plasma cells in the bone marrow greater than or equal to 10% or a documented clonal plasmacytoma (either by immuno-histochemistry or by Ig gene rearrangement), AND
* Presence of an M-component; an M-component (immunoglobulin G (IgG) or immunoglobulin A (IgA)) in serum greater than or equal to 1g/dl or in urine greater or equal to 200 mg/24 h.

ALTERNATIVELY, if the M-component criterion is not met:

* An abnormal serum free light chain (FLC) ratio on the serum FLC assay, or if the FLC ratio is normal,
* Baseline bone marrow must have 10% or greater clonal plasma cells

AND, IN ADDITION, presence of one or more of the following attributable to the disease (in the presence or absence of an M-component):

* Calcium elevation greater than 11.5 mg/dl (2.65 mmol/l)
* Renal insufficiency: serum creatinine greater than 2 mg/dl (177 mmol/l) or less than 60ml/min.
* Hemoglobin less than 10 g/dl (12.5 mmol/l) or 2 g/dl (1.25 mmol/l) below lower normal
* Bone disease (lytic lesions or osteopenia)
* Other evidence of disease activity: repeated infections, secondary amyloidosis, hyperviscosity, hypogammablobulinemia

Criteria for subjects with persistent or recurrent disease

Subjects with recurrent or persistent disease are eligible if:

* Criteria for initiating therapy for plasma cell myeloma (PCM) had been present at the time of initiation of therapy or there is clear clinical indication for salvage therapy.
* They have not undergone an autologous transplant for the treatment of PCM
* They have received no more than two salvage regimens for the treatment of recurrent or persistent PCM (each regimen may include more than one cycle)

Other eligibility criteria

-Age > 18 years and less than or equal to 75 years.

In subjects between 65 and 75 years of age, physiologic age and co-morbidity will be thoroughly evaluated before enrolling. Specifically, any history of cardiovascular pathology or symptoms not clearly fitting the exclusion criteria of Section 2.1.2 will prompt an evaluation by a Clinical Center Cardiologist and eligibility will be considered on a case-by-case basis.

* Karnofsky performance status of 70% or greater (Eastern Cooperative Oncology Group (ECOG) 0 or 1)
* Ejection fraction (EF) by multi-gated acquisition scan (MUGA) or 2-D echocardiogram within institution normal limits. In case of low ejection fraction (EF), the subject may remain eligible after a stress echocardiogram is performed if the EF is more than 35% and if the increase in EF with stress is estimated at 10% or more.
* creatinine clearance > 25ml/min (measured on a 24 hour urine collection)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3 x upper limit of normal
* Bilirubin less than or equal to1.5 (except if due to Gilbert's disease)
* Corrected carbon dioxide diffusing capacity (DLCO) greater than or equal to 40% on pulmonary function tests

EXCLUSION CRITERIA:

* Prior allogeneic or autologous stem cell transplantation
* Prior treatment with Carfilzomib (CFZ) is not an exclusion
* History of recent (< 6 months) cerebrovascular accident
* History of documented recent (< 6 months) pulmonary embolus
* Clinically significant cardiac pathology:
* Myocardial infarction within 6 months prior to enrollment,
* Class III or IV heart failure according to New York Heart Association (NYHA),
* Uncontrolled angina,
* Severe uncontrolled ventricular arrhythmias, or
* Electrocardiographic evidence of acute ischemia or active conduction abnormalities felt to pose a significant cardiac riks by a Cardiology consultant
* Patients with a history of coronary artery bypass grafting or angioplasty will receive a cardiology evaluation and be considered on a case-by-case basis.
* Human immunodeficiency virus (HIV) seropositive
* Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to enrollment
* Active hepatitis B or C infection
* Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment
* Major surgery within 21 days prior to enrollment
* Non-hematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
* Significant neuropathy (Grades 3 4, or Grade 2 with pain) within 14 days prior to randomization
* Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize CFZ)
* Patients known or found to be pregnant
* Female patients of childbearing age who are unwilling to practice contraception
* Patients may be excluded at the discretion of the principal investigator (PI) if it is deemed that allowing participation would represent an unacceptable medical or psychiatric risk.
* Patients must be able to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-07; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E Gress, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Rajkumar SV, Blood E, Vesole D, Fonseca R, Greipp PR; Eastern Cooperative Oncology Group. Phase III clinical trial of thalidomide plus dexamethasone compared with dexamethasone alone in newly diagnosed multiple myeloma: a clinical trial coordinated by the Eastern Cooperative Oncology Group. J Clin Oncol. 2006 Jan 20;24(3):431-6. doi: 10.1200/JCO.2005.03.0221. Epub 2005 Dec 19. PMID 16365178
- [Background] Tosi P, Zamagni E, Cellini C, Plasmati R, Cangini D, Tacchetti P, Perrone G, Pastorelli F, Tura S, Baccarani M, Cavo M. Neurological toxicity of long-term (>1 yr) thalidomide therapy in patients with multiple myeloma. Eur J Haematol. 2005 Mar;74(3):212-6. doi: 10.1111/j.1600-0609.2004.00382.x. PMID 15693790

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study did not progress to the phase II portion. The study was closed prematurely because the investigator left the National Institutes of Health.
Period: Overall Study
Arm/Group | Cohort 1- CFZ 20 mg/m^2 (Day 1,2) | Cohort 2- CFZ 20 mg/m^2 (Day 1,2,8,9) | Cohort 3-CFZ 20 mg/m^2 (Day1,2,8,9/AHCT)
Started | 3 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 2 | 0 | 0
Not completed — Principal Investigator discretion | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1- CFZ 20 mg/m^2 (Day 1,2) | Cohort 2- CFZ 20 mg/m^2 (Day 1,2,8,9) | Cohort 3-CFZ 20 mg/m^2 (Day1,2,8,9/AHCT) | Total
Number analyzed (Participants) | 3 | 0 | 0 | 3
Age, Categorical [Number; unit: participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 3 |  |  | 3
  >=65 years | 0 |  |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (10.39) |  |  | 49.6 (10.39)
Gender [Number; unit: participants]
  Female | 1 |  |  | 1
  Male | 2 |  |  | 2
Ethnicity (NIH/OMB) [Number; unit: participants]
  Hispanic or Latino | 0 |  |  | 0
  Not Hispanic or Latino | 3 |  |  | 3
  Unknown or Not Reported | 0 |  |  | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 |  |  | 0
  Asian | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  |  | 0
  Black or African American | 1 |  |  | 1
  White | 2 |  |  | 2
  More than one race | 0 |  |  | 0
  Unknown or Not Reported | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Engraftment Failure Transplant Related Mortality
Description: Engraftment failure is defined as the failure to achieve neutrophil engraftment by day 21; defined from day 0, day of autologous hematopoietic cell transplantation (AHCT), as the first of three consecutive days on which the patient's absolute neutrophil count is greater than 0.5x10(9)/l following the nadir. Transplant related mortality is defined as any subject who dies in the first 100 days post-AHCT of any non-relapse related cause.
Time Frame: up to day 100
Measure: Number; unit: participants
Arm/Group | Cohort 1- CFZ 20 mg/m^2 (Day 1,2) | Cohort 2- CFZ 20 mg/m^2 (Day 1,2,8,9) | Cohort 3-CFZ 20 mg/m^2 (Day1,2,8,9/AHCT)
Number analyzed (Participants) | 1 | 0 | 0
participants | 0 |  |

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 8 months and 15 days
Population: Analysis of dose limiting toxicities (DLTs) was planned but not performed due to study termination; this Outcome Measure captures any events that occurred.
Measure: Number; unit: participants
Arm/Group | Cohort 1- CFZ 20 mg/m^2 (Day 1,2) | Cohort 2- CFZ 20 mg/m^2 (Day 1,2,8,9) | Cohort 3-CFZ 20 mg/m^2 (Day1,2,8,9/AHCT)
Number analyzed (Participants) | 3 | 0 | 0
participants | 1 |  |

3. Secondary Outcome: Evaluate the Immune Reconstitution Post-Pre-autologous Hematopoietic Cell Transplantation (AHCT) Following Carfilzomib (CFZ) Therapy
Time Frame: Post-AHCT following CFZ therapy
Population: This outcome measure was not done because the study was closed prematurely because the investigator left the National Institutes of Health.
Groups:
- Cohort 1- CFZ 20 mg/m^2 (Day 1,2); Cohort 2- CFZ 20 mg/m^2 (Day 1,2,8,9); Cohort 3-CFZ 20 mg/m^2 (Day1,2,8,9/AHCT): Phase I/II study on the backbone of high-dose melphalan on day -2 pre-autologous hematopoietic cell transplantation (AHCT)
  •Addition of an increasing number of doses of Carfilzomib (CFZ) in the early post-AHCT period introduced in a step-wise fashion in 3 successive cohorts of 3 to 15 subjects:
  Cohort 1: add CFZ 20 mg/m^2 intravenous (IV) on days +1, +2
  Cohort 2 : add CFZ 20 mg/m^2 IV on days: +1, +2, +8, +9
  Cohort 3: add CFZ 20 mg/m^2 IV on days: +1, +2, +8, +9 and add an early post-AHCT consolidation following engraftment: CFZ 20 mg/m^2 IV given on days 42-43 then CFZ 56 mg/m^2 IV given on days 49-50, 56-57, then on days 70.
  Carfilzomib
  Melphalan
  Filgrastim
Arm/Group | Cohort 1- CFZ 20 mg/m^2 (Day 1,2) | Cohort 2- CFZ 20 mg/m^2 (Day 1,2,8,9) | Cohort 3-CFZ 20 mg/m^2 (Day1,2,8,9/AHCT)
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Evaluate the Effects of the Addition of Carfilzomib (CFZ) in the Early Post-Pre-autologous Hematopoietic Cell Transplantation (AHCT) Period on the Response Rate at Day 100 Post-AHCT
Time Frame: Day 100 post-AHCT
Population: as for outcome 3
Arm/Group | Cohort 1- CFZ 20 mg/m^2 (Day 1,2) | Cohort 2- CFZ 20 mg/m^2 (Day 1,2,8,9) | Cohort 3-CFZ 20 mg/m^2 (Day1,2,8,9/AHCT)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Cohort 1- CFZ 20 mg/m^2 (Day 1,2) | Cohort 2- CFZ 20 mg/m^2 (Day 1,2,8,9) | Cohort 3-CFZ 20 mg/m^2 (Day1,2,8,9/AHCT)
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/3 | 0/0 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1- CFZ 20 mg/m^2 (Day 1,2) (N=3) | Cohort 2- CFZ 20 mg/m^2 (Day 1,2,8,9) (N=0) | Cohort 3-CFZ 20 mg/m^2 (Day1,2,8,9/AHCT) (N=0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was closed prematurely because the investigator left the National Institutes of Health.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No